CLINICAL TRIAL: NCT00039455
Title: A Phase I Study of Herceptin/Flavopiridol in HER-2 Positive Metastatic Breast Cancer
Brief Title: Trastuzumab and Flavopiridol in Treating Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00035; 01-177; P50CA089393 (NIH); CDR0000069385 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Trastuzumab; alvocidib

ARMS (1):
- Treatment (trastuzumab and alvocidib) (Experimental): Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15 followed by flavopiridol IV continuously over 24 hours on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Drug: alvocidib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining trastuzumab with flavopiridol may kill more tumor cells. Phase I trial to study the effectiveness of combining trastuzumab with flavopiridol in treating patients who have metastatic breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of flavopiridol in combination with Herceptin in HER-2 positive metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To determine the dose of flavopiridol necessary to achieve a target plasma level of 300-500 nM of flavopiridol in combination with a fixed dose of Herceptin.

II. To assess the feasibility of measuring cyclin D1 in circulating tumor cells and tissue biopsies before and after therapy as a surrogate marker of flavopiridol activity.

III. To monitor target activity of flavopiridol and Herceptin in plasma, circulating tumor cells and tissue biopsies from breast cancer patients.

OUTLINE: This is a multicenter, dose-escalation study of flavopiridol.

Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15 followed by flavopiridol IV continuously over 24 hours on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose is determined (MTD). The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional cohort of 10 patients receives flavopiridol at the MTD and trastuzumab on the once weekly schedule to assess the true toxicity rate. A second cohort of 10 patients receives flavopiridol at the MTD and trastuzumab once every 21 days to assess the tolerability of this schedule.

PROJECTED ACCRUAL: A total of 30-50 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer, with stage IV disease; patients without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis by physical exam or radiologic study
* Either the primary tumor or the metastasis must overexpress HER2; acceptable methods of measurement of HER2 expression include immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH); tumors tested by IHC must be 3+ positive for HER2 overexpression using the DAKO Herceptest or the CB-11 antibody (recently FDA approved for HER-2 testing); tumors tested by FISH must be positive by either the Vysis Pathyvision method or the Ventana INFORM method; patients may have measurable or evaluable disease
* Patients may have received 0-3 prior chemotherapeutic regimens for metastatic breast cancer
* Patients may have received up to two prior Herceptin-containing regimens in the metastatic setting
* Patients may have received prior radiation therapy in either the metastatic or early stage settings; radiation therapy must be completed at least 7 days prior to study participation
* Patients may have received hormonal therapy (therapies) in the adjuvant or metastatic setting; patients must discontinue hormonal therapy prior to study participation
* Life expectancy of greater than 6 months
* ECOG performance status < 2 (Karnofsky > 60%)
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 mg/dl
* AST(SGOT)/ALT(SGPT) =< 3 X upper limit normal
* Creatinine =< 2.0 mg/dl
* LVEF >= 50%
* EKG no acute changes
* Patients may not receive concurrent hormonal therapy, chemotherapy, or radiation treatments while on study; patients requiring radiation therapy during protocol-based treatment will be taken off study with the exception of whole brain radiation or stereotactic radiosurgery for brain metastases; protocol-based therapy will be held during the therapy and for 1 week after treatment but may be resumed; patients may not receive other experimental treatments while on study; patient receiving bisphosphonates may continue to receive treatment while on study; patients may initiate bisphosphonate therapy while on study provided that there has been no evidence of progressive disease and that the bone sites do not constitute the only sites of evaluable disease; if patients are on Lupron prior to the start of this trial, than they must continue on Lupron throughout the course of this study
* Patients must be neither pregnant nor expect becoming pregnant or conceiving a child while on study; women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had more than three chemotherapy regimens in the metastatic setting, more than two Herceptin-containing regimens in the metastatic setting, radiation therapy within 1 week prior to study entry, or those who have not recovered from reversible adverse events due to prior treatments for cancer, are ineligible
* Patients with active brain metastases or leptomengingeal carcinomatosis are excluded from this clinical trial; patients with a history of treated CNS metastases are eligible if they do not have active symptoms from their CNS disease
* Patients with a history of grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in the study are ineligible; patients who experienced grade 1 or 2 hypersensitivity reactions to prior Herceptin are eligible IF these reactions did not prevent further administration
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are ineligible
* Pregnant women are excluded from this study
* Patients with a contraindication to taking coumadin or other warfarin products are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-04; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT) assessed using National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 2.0 | 3 weeks

SECONDARY OUTCOMES:
Measures of circulating extracellular domain of HER-2 in plasma | Up to 3 years
  Descriptive analyses will be performed.
Measures of HER-2, Cyclin D1 and activated Rb in circulating tumor cells | Up to 3 years
  Descriptive analyses will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsay Harris, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States